CLINICAL TRIAL: NCT01752569
Title: Phase I/II Study of Oral MEK Inhibitor Selumetinib (AZD6244 Hyd-Sulphate) in Combination With Highly Active Anti-Retroviral Therapy (HAART) in AIDS-associated Kaposi's Sarcoma (KS).
Brief Title: A Study of Selumetinib in Patients With Kaposi's Sarcoma
Acronym: SCART
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Birmingham (Other); AstraZeneca (Industry); Thermo Fisher Scientific, Inc (Industry); Cancer Research UK (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH16059; 2011-003099-35 (EudraCT Number)
Record Dates: First submitted 2012-08-17; First posted 2012-12-19 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: AIDS-related Kaposi's Sarcoma
Keywords: HIV; Kaposi's sarcoma; Anti-retroviral therapy; HAART; AIDS
MeSH Terms: conditions — AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Selumetinib treatment (Experimental): Phase I is a dose-finding study to discover the maximum tolerated dose of selumetinib in combination with HAART. Phase II will consider the efficacy of selumetinib for treating Kaposi's sarcoma at the recommended phase II dose discovered in phase I.
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — The treatment schedule requires selumetinib to be taken either once daily at the same time each day or twice daily approximately 12 hours apart. Selumetinib should be taken with water at least 2 hours after a meal and 1 hour before the next meal. Selumetinib capsules will be administered in a continuous 21 day cycle (6 cycles), unless disease progression occurs.
  For phase I there were 4 potential dosing levels:
  Level -1 - 50mg once daily (od) (50mg daily total)
  Level 1 (starting dose level for phase I) - 50mg bi-daily (bd) (100mg daily total)
  Level 2 - 75mg bd (150mg daily total)
  Level 3 - 100mg bd (200mg daily total)
  Phase I has been completed and identified 75mg bd as the recommended phase II dose.
  Phase II has begun and is utilising a dose of 75mg bd of selumetinib.
  Other Names: AZD6244

SUMMARY:
Cancer is a leading cause of death in individuals living with human immunodeficiency virus (HIV), and Kaposi's sarcoma (KS) remains the commonest HIV-associated cancer. KS is caused when individuals become infected with both HIV and another virus, Human herpesvirus-8 (HHV-8). Laboratory studies have shown that HHV-8 can stimulate biological pathways within KS lesions which promotes their growth. Selumetinib targets these pathways and may therefore be a useful new therapy for KS. Phase I of this trial aims to identify the best dose for the use of selumetinib and investigate the effects of selumetinib treatment on the anti-viral treatment HIV patients receive to control HIV infection. Phase II of this trial will investigate how well selumetinib works as a treatment for KS at the best dose determined in phase I.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

HIV AND KS

The prevalence of HIV in the United Kingdom (UK) is rising with about 83,000 living with HIV and 7,000 new cases per annum (pa). At diagnosis a third of patients have severe immune-suppression with a cluster of differentiation 4 (CD4) positive cell count less than 200/mm3 (HPA, 2009), which is associated with opportunistic infections and an increase in various tumours. Cancer is a leading cause of death in individuals living with HIV, and KS remains the commonest AIDS-associated malignancy. In a UK prospective cohort followed in the Highly Active Anti-Retroviral Therapy (HAART) era, 5.5% of HIV positive patients developed KS (Stebbing et al., 2006).

KS is associated with co-infection with HIV and human herpesvirus-8 (HHV-8). Patients typically present with multi-focal cutaneous disease often with associated lymphoedema. Extra-cutaneous disease commonly involves the gastrointestinal tract, lung, liver and spleen. For early KS, initiation of HAART may be sufficient to control the disease and radiotherapy is of benefit for localised disease (Di Lorenzo et al., 2007). Currently the only alternative for progressive localised disease is cytotoxic chemotherapy.

Cytotoxic chemotherapy with liposomal anthracycline or taxanes, is indicated in patients with widespread cutaneous KS, extensive oral disease or symptomatic visceral involvement (Bower et al., 2008). Pegylated liposomal doxorubicin (PLD) 20mg/m2 q 3 weeks as first-line therapy in combination with HAART is reported to give tumour response in 55% of patients and median progression free survival (PFS) of 22 weeks (Cooley et al., 2007). Second-line therapy with low dose paclitaxel (100mg/m2 q 2 weeks) is reported to give a response rate of 56% with median PFS of 39 weeks (Tulpule et al., 2002). However the majority of patients' progress despite chemotherapy and new treatment alternatives are required.

JUSTIFICATION FOR DESIGN

Selumetinib has been tested in a number of phase I and phase II trials as both monotherapy and combined with cytotoxic chemotherapy in patients with advanced solid malignancies. A toxicity profile and recommended dose has been established in these patients. Selumetinib has not been tested in combination with HAART. No significant interactions are predicted between Selumetinib and HAART however a phase I study is required to investigate the pharmacokinetic effects of combining these drugs. In particular we wish to establish that Selumetinib will not reduce the efficacy of HAART.

This trial is an open-label multi-centre phase I/II study to investigate the use of selumetinib as a potential treatment for HIV-associated KS. Phase I is an accelerated dose finding study with dosing commencing at 1 dose level below that recommended for monotherapy or in combination with cytotoxic chemotherapy. The aims of phase I are to identify a maximum tolerated dose (MTD) for selumetinib in patients on HAART whilst proving selumetinib does not reduce the efficacy of HAART. Phase II aims to provide evidence of the efficacy of selumetinib as a treatment for KS. Evidence of efficacy will be assessed via objective response rate to treatment and will be used to develop a protocol for a future randomised phase II/III study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed KS.
* Measurable disease according to ACTG criteria.
* Evidence of disease progression in the past 6 months. No anti-cancer treatment within one month prior to commencing trial treatment.
* Progressive cutaneous or nodal KS not requiring chemotherapy OR progressive KS following cytotoxic chemotherapy.
* Adequate haematological function:

  * Haemoglobin ≥ 9 g/dL
  * Absolute neutrophil count ≥ 1.5 x 10 9/L
  * Platelets ≥ 100 x 10 9/L
* Adequate hepatic function:

  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN), except if the patient is established on the anti-retroviral drug atazanavir (no upper limit) and has aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 x ULN
  * ALT ≤ 2.5 x ULN
  * AST ≤ 2.5 x ULN
* Adequate renal function:

  * Serum creatinine clearance > 50 ml/min (Cockcroft-Gault formula or 24 hour urine collection).
* Left ventricular function >50% normal
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* For selumetinib, women of child bearing age and child bearing potential MUST have a negative pregnancy test prior to study entry AND be using an adequate contraception method, which must be continued while on treatment and for at least 4 weeks after the study treatment has ended.
* Male patients must agree to use an effective contraception method while on treatment and for at least 16 weeks after the study treatment has ended (barrier contraception is recommended for all individuals living with HIV).
* Written informed consent

Exclusion Criteria:

* HIV viral load > 200 copies/ml.
* Any previous treatment with a Ras, Raf or MEK inhibitor.
* Active opportunistic infections.
* Known hepatitis B, hepatitis C.
* Clinical evidence of uncontrolled hypertension (systolic BP > 150 mmHg or diastolic BP > 90 mmHg on 2 readings ≥ 1 hour apart).
* Clinical evidence of heart failure (New York Heart Association ≥Class II).
* Clinical evidence of atrial fibrillation (heart rate > 100 bpm) or unstable ischaemic heart disease (MI within 6 months prior to starting treatment or angina requiring the use of nitrates > once weekly).
* Major surgery within 4 weeks prior to starting selumetinib.
* Evidence of any psychological, familial, sociological or geographical condition potentially hampering protocol compliance.
* Clinical judgement by the Investigator that the patient should not participate in the study.
* Refractory nausea, vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease) or significant bowel resection that would preclude adequate absorption.
* Treatment with any investigational product within 28 days of registration
* Pregnant or breast-feeding women.
* Japanese ethnicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Toxicity of Selumetinib in Combination with HAART | 3.5 years
  The primary objective of phase I of this study is to identify a safe dose for Selumetinib in combination with HAART (called the recommended phase II dose) for use in an expanded phase II cohort. The recommended phase II dose will be elucidated using a dose-escalation algorithm which will be used to allocate patients to cohorts at a given dose level or expand the numbers of patients allocated to a given dose level dependent on the previous occurrence of specifically pre-defined toxicities (according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0) called dose limiting toxicities. Dose limiting toxicities will only be recorded in phase I to obtain a recommended phase II dose. However, all toxicities/adverse events will be recorded throughout both phase I and II of the trial according to CTCAE version 4.0.
Objective Response Rate to Selumetinib Treatment | 3.5 years
  Objective response rate to treatment will be assessed using the AIDS Clinical Trials Group (ACTG) Oncology Committee Documentation of Disease and Definition of Response criteria. This will be the primary measure of efficacy to test the null hypothesis that the recommended phase II dose will produce an objective response in less than 10% of patients. The alternative hypothesis that the recommended phase II dose will produce an objective response in more than 30% of patients will also be tested.

SECONDARY OUTCOMES:
Peripheral Blood Mononuclear Cell (PBMC) Sub-study | 3.5 years
  Effects of selumetinib treatment on PBMCs will be assessed by isolating these cells and subjecting them to the following analyses: -
  * Levels of pERK, downstream targets c-fos and c-myc and key apoptotic proteins Bad and Bcl-2 will be assessed by Western blotting of lysed viable PBMCs.
  * PBMCs will be challenged with Toll-like Receptor (TLR) 4 and 9 agonists and production of Interleukins (ILs) including IL-1β, IL-6, IL-10 and IL-12 alongside type 1 interferon and tumor necrosis factor alpha (TNFα) will be measured by cytometric bead array of culture supernatants.
  * PBMC reactive oxygen species production and cell survival assessment will be measured flow cytometry.
Number of Completed Cycles | 3.5 years
  Upon patients discontinuing trial treatment, the number of cycles of Selumetinib treatment in combination with HAART that patients received will be recorded.
HIV Viral Load and CD4 Count | 3.5 years
  HIV control will be monitored through assessment of HIV-1 viral load and CD4 cell counts throughout the trial.
HAART Drug Levels | 2 years
  HAART drug pharmacokinetics will be assessed to discover the effects of selumetinib on HAART drug metabolism (during phase I only).
Selumetinib and Metabolite Serum Levels | 2 years
  The pharmacokinetics of selumetinib and its metabolites will be assessed to discover the effects of HAART on selumetinib metabolism (during phase I only).
Serum Angiogenic Biomarkers Levels | 3.5 years
  Pharmacodynamic effects of Selumetinib in combination with HAART will be assessed by: -
  * Quantification of serum concentrations of angiogenic markers including serum Angiopoietin 2 (Ang-2), IL-6 and Vascular Endothelial Growth Factor (VEGF) as analysed via Enzyme-Linked Immunosorbent Assay (ELISA).
  * Analysis of tissue biopsies for pERK levels in tumour tissues and other downstream markers including c-fos, c-myc, apoptotic markers (e.g. Bad and Bcl-2) and for adaptive changes in Phosphoinositide 3-kinase (PI3K), Akt and other Mitogen-Activated Protein Kinase (MAPK) pathways such as c-Jun N-terminal kinase (JNK) and p38.
Progression Free Survival | 3.5 years
  Progression free survival will be assessed for 6 months from commencing selumetinib treatment for each patient using ACTG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bower, Professor, Principal Investigator — Chelsea & Westminster Hospital, London; Diana Ritchie, Dr., Principal Investigator — Beatson West of Scotland Cancer Centre, Glasgow; Sarah Westwell, Dr., Principal Investigator — Royal Sussex County Hospital, Brighton; Michael Leahy, Dr, Principal Investigator — The Christie Hospital, Manchester; Robin Young, Dr, Principal Investigator — West Park Hospital, Sheffield; Grant Stewart, Dr, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Brighton and Sussex University Hospitals, Brighton
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital, London
  - Chelsea & Westminster Hospital, London
  - The Christie Hospital, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- [Background] Adjei AA, Cohen RB, Franklin W, Morris C, Wilson D, Molina JR, Hanson LJ, Gore L, Chow L, Leong S, Maloney L, Gordon G, Simmons H, Marlow A, Litwiler K, Brown S, Poch G, Kane K, Haney J, Eckhardt SG. Phase I pharmacokinetic and pharmacodynamic study of the oral, small-molecule mitogen-activated protein kinase kinase 1/2 inhibitor AZD6244 (ARRY-142886) in patients with advanced cancers. J Clin Oncol. 2008 May 1;26(13):2139-46. doi: 10.1200/JCO.2007.14.4956. Epub 2008 Apr 7. PMID 18390968
- [Background] Banerji U, Camidge DR, Verheul HM, Agarwal R, Sarker D, Kaye SB, Desar IM, Timmer-Bonte JN, Eckhardt SG, Lewis KD, Brown KH, Cantarini MV, Morris C, George SM, Smith PD, van Herpen CM. The first-in-human study of the hydrogen sulfate (Hyd-sulfate) capsule of the MEK1/2 inhibitor AZD6244 (ARRY-142886): a phase I open-label multicenter trial in patients with advanced cancer. Clin Cancer Res. 2010 Mar 1;16(5):1613-23. doi: 10.1158/1078-0432.CCR-09-2483. Epub 2010 Feb 23. PMID 20179232
- [Background] Bodoky G, Timcheva C, Spigel DR, La Stella PJ, Ciuleanu TE, Pover G, Tebbutt NC. A phase II open-label randomized study to assess the efficacy and safety of selumetinib (AZD6244 [ARRY-142886]) versus capecitabine in patients with advanced or metastatic pancreatic cancer who have failed first-line gemcitabine therapy. Invest New Drugs. 2012 Jun;30(3):1216-23. doi: 10.1007/s10637-011-9687-4. Epub 2011 May 19. PMID 21594619
- [Background] Bower M, Collins S, Cottrill C, Cwynarski K, Montoto S, Nelson M, Nwokolo N, Powles T, Stebbing J, Wales N, Webb A; AIDS Malignancy Subcommittee. British HIV Association guidelines for HIV-associated malignancies 2008. HIV Med. 2008 Jul;9(6):336-88. doi: 10.1111/j.1468-1293.2008.00608.x. No abstract available. PMID 18705759
- [Background] Cooley T, Henry D, Tonda M, Sun S, O'Connell M, Rackoff W. A randomized, double-blind study of pegylated liposomal doxorubicin for the treatment of AIDS-related Kaposi's sarcoma. Oncologist. 2007 Jan;12(1):114-23. doi: 10.1634/theoncologist.12-1-114. PMID 17227906
- [Background] Di Lorenzo G, Konstantinopoulos PA, Pantanowitz L, Di Trolio R, De Placido S, Dezube BJ. Management of AIDS-related Kaposi's sarcoma. Lancet Oncol. 2007 Feb;8(2):167-76. doi: 10.1016/S1470-2045(07)70036-0. PMID 17267331
- [Background] Krown SE, Metroka C, Wernz JC. Kaposi's sarcoma in the acquired immune deficiency syndrome: a proposal for uniform evaluation, response, and staging criteria. AIDS Clinical Trials Group Oncology Committee. J Clin Oncol. 1989 Sep;7(9):1201-7. doi: 10.1200/JCO.1989.7.9.1201. PMID 2671281
- [Background] Sharma-Walia N, Krishnan HH, Naranatt PP, Zeng L, Smith MS, Chandran B. ERK1/2 and MEK1/2 induced by Kaposi's sarcoma-associated herpesvirus (human herpesvirus 8) early during infection of target cells are essential for expression of viral genes and for establishment of infection. J Virol. 2005 Aug;79(16):10308-29. doi: 10.1128/JVI.79.16.10308-10329.2005. PMID 16051824
- [Background] Stebbing J, Sanitt A, Nelson M, Powles T, Gazzard B, Bower M. A prognostic index for AIDS-associated Kaposi's sarcoma in the era of highly active antiretroviral therapy. Lancet. 2006 May 6;367(9521):1495-502. doi: 10.1016/S0140-6736(06)68649-2. PMID 16679162
- [Background] Tulpule A, Groopman J, Saville MW, Harrington W Jr, Friedman-Kien A, Espina BM, Garces C, Mantelle L, Mettinger K, Scadden DT, Gill PS. Multicenter trial of low-dose paclitaxel in patients with advanced AIDS-related Kaposi sarcoma. Cancer. 2002 Jul 1;95(1):147-54. doi: 10.1002/cncr.10634. PMID 12115328
- [Background] Vart RJ, Nikitenko LL, Lagos D, Trotter MW, Cannon M, Bourboulia D, Gratrix F, Takeuchi Y, Boshoff C. Kaposi's sarcoma-associated herpesvirus-encoded interleukin-6 and G-protein-coupled receptor regulate angiopoietin-2 expression in lymphatic endothelial cells. Cancer Res. 2007 May 1;67(9):4042-51. doi: 10.1158/0008-5472.CAN-06-3321. PMID 17483315
- [Background] Wang HW, Trotter MW, Lagos D, Bourboulia D, Henderson S, Makinen T, Elliman S, Flanagan AM, Alitalo K, Boshoff C. Kaposi sarcoma herpesvirus-induced cellular reprogramming contributes to the lymphatic endothelial gene expression in Kaposi sarcoma. Nat Genet. 2004 Jul;36(7):687-93. doi: 10.1038/ng1384. Epub 2004 Jun 27. PMID 15220918
- [Background] Xie J, Ajibade AO, Ye F, Kuhne K, Gao SJ. Reactivation of Kaposi's sarcoma-associated herpesvirus from latency requires MEK/ERK, JNK and p38 multiple mitogen-activated protein kinase pathways. Virology. 2008 Feb 5;371(1):139-54. doi: 10.1016/j.virol.2007.09.040. Epub 2007 Oct 26. PMID 17964626
- [Background] Yang X, Gabuzda D. Regulation of human immunodeficiency virus type 1 infectivity by the ERK mitogen-activated protein kinase signaling pathway. J Virol. 1999 Apr;73(4):3460-6. doi: 10.1128/JVI.73.4.3460-3466.1999. PMID 10074203
- See also: Health Protection Agency "HIV in the United Kingdom" Report 2009 — http://www.hpa.org.uk